CLINICAL TRIAL: NCT00040495
Title: An Efficacy and Safety Study of Intravenous Pantoprazole in the Prevention of Recurrent Peptic Ulcer Bleeding After Successful Hemostasis
Brief Title: Study Evaluating Pantoprazole in Peptic Ulcer Hemorrhage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: 3001K2-315
Record Dates: First submitted 2002-06-26; First posted 2002-06-28 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic; Ulcer; Hemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Ulcer; Hemorrhage | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of intravenous pantoprazole in the prevention of rebleeding in patients with bleeding peptic ulcer disease after successful endoscopic hemostatic therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be men or non-pregnant women at least 18 years of age
* Patients who present with a gastric or duodenal ulcer

Exclusion Criteria:

* Patients with ulcer appearance of clean base (non-oozing, non-spurting) or flat pigmented spot; adherent clots not removed by irrigation
* Patients presenting with active bleeding and/or NBVV at 2 or more separate sites
* Patients with any severe concomitant diseases, eg, end stage liver or renal disease, or unstable cardiovascular, pulmonary, renal, hepatic, or gastrointestinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2001-04; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer